CLINICAL TRIAL: NCT02940197
Title: Comparison of the Effect of MediterrAsian Diet With Two Different Calorie Restriction on Anthropometric Indices in Carriers of FTO rs9939609 Polymorphism With Overweigh: Toward Personalized Nutrition
Brief Title: Comparison of Two Calorie Restricted MediterrAsian Diet on Weight Loss in FTO rs9939609 Overweight Carriers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mahsa Mehrdad, Ph.D Candidate, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ir.sums.rec.1395.100
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2017-09

CONDITIONS: Obesity; Dietary Modification
Keywords: overweight; Caloric Restriction
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- restricted diet (Experimental): Mediterrasian diet according to adjusted ideal body weight with 500 calorie restriction
  Interventions: Behavioral: MediterrAsian diet
- Non restricted diet (Experimental): Mediterrasian diet according to adjusted ideal body weight without 500 calorie restriction
  Interventions: Behavioral: MediterrAsian diet

INTERVENTIONS:
Behavioral: MediterrAsian diet — no other description

SUMMARY:
Background: Obesity treatment should be individualized since some calorie restricted diet doesn't work for some individuals.

Objective: we assess the effect of two different calorie restriction with MediterrAsian diet on weight loss of FTO rs9939609 carriers with overweight.

Methods: we recruit 80 healthy overweight participants aged 20-45 years that randomly allocated in two interventional group [group 1: Mediterrasian diet according to adjusted ideal body weight with 500 calories restriction (RD) and group 2: without 500 calories restriction (NRD)+ Moderate physical activity]. Anthropometric indices will be assesses for all participants weekly for two month. The criteria for weight loss is 250-500 grams weekly. Metabolic indices, physical activity and psychologic aspects will be assesses at baseline and the end of the intervention. Dietary adherence will be checked by 24hr recalls at day 0, 30 and 60. At the end of the study, we compare carriers with different alleles (AA+TA and TT) in two intervention groups to find out which calorie restriction is appropriate for each genotype. Significant p-value is less than 0.05.

DETAILED DESCRIPTION:
no data yet

ELIGIBILITY:
Minimum age: 20 years Maximum age: 45 years Gender: Both Accepts Healthy Volunteers?: Yes

Criteria: Inclusion Criteria:

* BMI range: 24.9-29.9 (overweight)
* Ethnicity: Persian

Exclusion Criteria:

* History of any metabolic diseases like Diabetes, CVD, Thyroid problems and ... .
* History of depression
* Pregnancy, trying to become pregnant or breast feeding
* Smoking
* Use of alcohol
* Significant weight loos during last two months (>5 kilograms)
* being on a diet during last two months
* Use of any drug or supplement

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
weight loss | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz university of medical sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Undecided